CLINICAL TRIAL: NCT03971006
Title: Immune Alveolar Alterations During Pneumonia-Associated Acute Respiratory Distress Syndrome
Acronym: PICARD2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 190092
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute respiratory distress syndrome (ARDS); Pneumonia; Septic Shock; bronchoalveolar lavage
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchoalveolar lavage fluid and blood samples (2 heparinized tubes (8 ml) for performing functional tests in the blood compartment and 1 dry 4 ml tube for subsequent cytokine assay (Luminex® analysis) on serum) will be collected in ARDS patients within 48 hours of intubation and in controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Immunocompetent ARDS patients: (n=50) Patients with moderate-to-severe pneumonia-associated Acute Respiratory Distress Syndorme (ARDS) and no immunosuppression (excluding patients with HIV infection, solid tumor or hematological malignancies, organ transplant or taking steroids since more than 4 weeks).
- Immunosuppressed ARDS patients: (n=50) Patients with moderate-to-severe pneumonia-associated Acute Respiratory Distress Syndorme (ARDS) (Berlin definition (2)) and previously known immunosuppression (as listed above). These patients will allow comparing the cell defects observed in the study population to those observed in immunosuppressed patients.
- Controls: (n=10) Patients undergoing a bronchoscopy with Bronchoalveolar Liquid (BAL) as part of routine care but having neither ARDS nor active lung infection, infiltrating lung disease or immunosuppression. These patients will allow quantifying normal levels of the studied biomarkers in the alveolar and blood compartments.

SUMMARY:
Sepsis is a dysregulated host response to severe life-threatening infections, leading to organ failure and death in up to 40% of patients with septic shock. Pulmonary infections are the main cause of community-acquired sepsis and frequently lead to the development of acute respiratory distress syndrome(ARDS). Features of immunosuppression, including diminished cell surface monocyte human leukocyte antigen DR (mHLA-DR) expression, are strongly associated with hospital mortality. Such decrease in HLA-DR expression on antigen-presenting cells has been associated with impairment of microbial antigens to Tcells. Septic patients also show elevated expression of inhibitory receptors associated with cell exhaustion.. Yet, biochemical, flow cytometric and immunohistochemical findings consistent with immunosuppression have been observed in lungs and spleen of patients died of sepsis and multiple organ failure, demonstrating the relevance of studying these defects directly in organ tissues. A novel approach aimed to characterize the role and prognostic value of alveolar biomarkers measured directly in the injured lungs is warranted and supported by: -disappointing results of previous clinical trials attempting to restore the level of biomarkers measured on circulating cells; -evidences of regional immunosuppression in lungs of ARDS patients; -lung is the main site of hospital-acquired infections with a prevalence of ventilator-associated pneumonia in 30% over the course of Intensive Care Unit(ICU) stay in ARDS patients.

Investigators speculate that biomarkers measured on alveolar leukocytes (AL) surface, are important predictors of outcome and potential therapeutic targets in ICU patients with pneumonia-associated ARDS.

Investigators aim to explore whether biomarkers measured directly on AL from patients with pneumonia-associated ARDS are associated to regional pulmonary immunosuppression using leukocyte functional tests; and predictors of outcomes.

Bronchoalveolar lavage fluid(BALF) and blood samples will be collected in ARDS patients. Leukocyte populations and cell membrane biomarkers will be quantified using flow cytometry. Leukocyte functional tests will be performed ex vivo on leukocytes collected from BALF and blood samples. Pharmacological interventions will be performed ex vivo.

This project aims to identify biomarkers associated with outcomes and potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Affiliated to a social security system
* Patient informed and have given his non opposition verbally (trustworthy or a family member non opposition is required if the patient is unable to give his non opposition)

Groupe 1 :

- Patient with ARDS secondary to pneumonia defined by following criteria: Intubation and mechanical ventilation for less than 48 hours Lung infection evolving since less than 7 days Bilateral pulmonary radiological opacities compatible with edema pulmonary lesion PaO2 / FiO2 ratio ≤ 300 mmHg with a positive expiratory pressure level ≥ 5 cmH2O

- Absence of immunosuppression (No HIV infection, bone marrow or solid organ transplantation, post-chemotherapy aplasia, immunosuppressive therapy or corticosteroid therapy (>200 mg / day of hydrocortisone or equivalent in the 4 weeks prior to inclusion))

Group 2 - Patient with ARDS secondary to pneumonia defined by following criteria: Intubation and mechanical ventilation for less than 48 hours Lung infection evolving since less than 7 days Bilateral pulmonary radiological opacities compatible with edema pulmonary lesion PaO2 / FiO2 ratio ≤ 300 mmHg with a positive expiratory pressure level ≥ 5 cmH2O

- Previously known immunosuppression (patient with HIV, solid tumor, solid organ transplantation or under corticosteroids therapy since at least 4 weeks before inclusion)

Group 3

* LBA indicated in usual care
* Absence of ARDS
* Absence of evolutionary infection
* Absence of infiltrative lung disease
* Absence of immunosuppression (No HIV infection, bone marrow or solid organ transplantation, post-chemotherapy aplasia, immunosuppressive therapy, corticosteroid therapy (> 200 mg / day of hydrocortisone or equivalent in the 4 weeks prior to inclusion))

Exclusion Criteria:

* Chronic respiratory insufficiency treated by long-term oxygen therapy and / or long-term respiratory assistance
* Child-Pugh C cirrhosis
* Pulmonary fibrosis
* Active lymphoid and myeloid malignant hemopathies
* Neutropenia (neutrophils <1500 / mm3)
* Patient moribund the day of inclusion or having an IGS II score greater than 90
* Irreversible neurological pathology: cerebral involvement, encephalic death
* Decision to limit active therapies
* Deep hypoxemia (PaO2 / FiO2 <75 mmHg)
* Patient protected by law
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1 : Immunocompetent Acute Respiratory Distress Syndorme (ARDS) patients Group 2 : Immunosuppressed ARDS patients Group 3 : Controls (no ARDS)
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-06-04 (Estimated); Study Completion 2022-06-28 (Estimated)

PRIMARY OUTCOMES:
HLA-DR expression level of alveolar monocytes at the early phase of infectious Acute Respiratory Distress Syndrome (ARDS) | at day 1 to day 3
  Measurement by flow cytometry phagocytosis and TNF-α synthesis of alveolar monocytes in immunocompetent patients, compared to immunocompromised patients

SECONDARY OUTCOMES:
Impact of the level of expression of PD-1 by alveolar CD8 + lymphocytes on their function during septic ARDS in immunocompetent and immunocompromised patients. | at day 1 to day 3
  Level of expression of PD-1 by alveolar CD8+ lymphocytes
Comparaison of the level of HLA-DR expression of alveolar monocytes between immunocompetent and immunosuppressed patients being managed for septic ARDS. | at day 1 to day 3
  Level of HLA-DR expression of alveolar monocytes
Link between the alveolar monocyte HLA-DR expression level and the prognosis of immunocompetent and immunosuppressed patients being managed for septic ARDS. | day 28
  Number of days without complication
Determine wether alveolar biomarkers (HLA-DR and PD-1) are potential candidates for immunomodulation | at day 1 to day 3
  To determine if the level of expression of HLA-DR and PD-1 can be modulated by pharmacological intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DE PROST, Principal Investigator — Assistance Publique Hôpitaux de Paris - CHU Henri Mondor - Créteil

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION